CLINICAL TRIAL: NCT00388401
Title: A Multicenter Phase III, Double-Blind, Placebo-Controlled, Parallel Study of ADL-8-2698 in Opioid-Induced Postoperative Bowel Dysfunction/Postoperative Ileus
Brief Title: Study of Alvimopan for the Management of Opioid-induced Postoperative Bowel Dysfunction/Postoperative Ileus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14CL313
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2008-10

CONDITIONS: Ileus
Keywords: Postoperative Ileus
MeSH Terms: conditions — Ileus | interventions — alvimopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alvimopan

SUMMARY:
Patients undergoing major abdominal surgery are at highest risk for developing postoperative ileus (POI), occurring in nearly all cases. Signs and symptoms of POI may include abdominal distention, bloating, persistent abdominal pain; nausea and/or vomiting; delayed passage or inability to pass flatus or stool; and inability to tolerate a solid diet. This study will test the ability of alvimopan 6 mg or 12 mg given 2 hours before the scheduled start of surgery to hasten the recovery of GI function in patients undergoing major abdominal surgery (bowel resection or abdominal hysterectomy).

DETAILED DESCRIPTION:
Postoperative ileus (POI) is temporary slowing down or stopping of bowel function and a slowing down of movement of contents of the intestines. This functional impairment persists for a variable duration following surgery, usually resolving within 1 day in the small intestine, 1 to 3 days in the stomach and 3 to 5 days in the colon. When POI persists for more than 5 days, it is generally considered severe, sometimes referred to as complicated or prolonged POI, and increases the risk for related morbidity. No drug therapy has been shown to consistently shorten the duration of POI. This study is designed to demonstrate that alvimopan, a novel, peripherally acting mu opioid receptor antagonist, accelerates the recovery of GI function in patients undergoing bowel resection of hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for a partial small/large bowel resection of primary anastomosis or total abdominal hysterectomy (simple or radical) via laparotomy
* Subject is scheduled to receive primary postoperative pain management with intravenous (i.v.) patient-controlled analgesia (PCA) opioids

Exclusion Criteria:

* Subject is scheduled for a total colectomy, colostomy, ileostomy
* Subject has complete bowel obstruction
* Subject is currently taking opioid analgesics or has taken opioid analgesics within the prior 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510
Dates: Start 2002-01; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
acceleration of gastrointestinal recovery

SECONDARY OUTCOMES:
time until ready for discharge based upon recovery of GI function
severity of GI symptoms
pain
opioid consumption
time to tolerate solid food
need for reinsertion of nasogastric tube
time until discharge order is written

CONTACTS AND LOCATIONS:
Overall Officials: Adolor Corporation, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (1):
- Adolor Corporation, Exton, Pennsylvania, United States

REFERENCES:
- [Result] Wolff BG, Michelassi F, Gerkin TM, Techner L, Gabriel K, Du W, Wallin BA; Alvimopan Postoperative Ileus Study Group. Alvimopan, a novel, peripherally acting mu opioid antagonist: results of a multicenter, randomized, double-blind, placebo-controlled, phase III trial of major abdominal surgery and postoperative ileus. Ann Surg. 2004 Oct;240(4):728-34; discussion 734-5. doi: 10.1097/01.sla.0000141158.27977.66. PMID 15383800
- [Derived] Ludwig K, Viscusi ER, Wolff BG, Delaney CP, Senagore A, Techner L. Alvimopan for the management of postoperative ileus after bowel resection: characterization of clinical benefit by pooled responder analysis. World J Surg. 2010 Sep;34(9):2185-90. doi: 10.1007/s00268-010-0635-9. PMID 20526599